CLINICAL TRIAL: NCT02211560
Title: A, Multi-center, Double-blind, Randomized, Placebo-controlled Study for the Efficacy of Phosphatidylserine in Mild Cognitive Impairment (MCI)
Brief Title: Investigating a Phosphatidylserine Based Dietary Approach for the Management of Mild Cognitive Impairment
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to difficulties in patient recruitment
Sponsor: Enzymotec (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: Vayacog_002
Record Dates: First submitted 2014-08-06; First posted 2014-08-07 (Estimated); Last update posted 2018-02-05 (Actual); Status verified 2018-02

CONDITIONS: Mild Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Phosphatidylserines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Identical looking cellulose capsules
  Interventions: Other: Placebo
- Phosphatidylserine (Experimental): Phosphatidylserine-omega-3, DHA enriched
  Interventions: Other: Phosphatidylserine

INTERVENTIONS:
Other: Phosphatidylserine
  Arms: Phosphatidylserine
Other: Placebo
  Arms: Placebo

SUMMARY:
The primary objective is to evaluate the efficacy and safety of phosphatidylserine (PS) on cognitive abilities in MCI

ELIGIBILITY:
Inclusion Criteria:

1. Age greater than or equal to 65 and less than or equal to 85 years.
2. Formal education greater than or equal to 10 years.
3. Male or female with a diagnosis of Mild Cognitive Impairment (MCI) 3. Male or female with a diagnosis of Mild Cognitive Impairment (MCI) as defined by Peterson, according to The following:

   3.1 Clinical Dementia Rating Scale total score (CDR) ≤0.5, and score of each one of the six categories ("box scores") ≤ 1. 3.2 Mini Mental State Exam > 24 3.3 Verbal Paired-Associated Learning test score according to the following ages: Ages 65-70 less than or equal to 18 Ages 71-85* less than or equal to 17

   *Eligibility of subjects aged between 70 and 71 (i.e., 70.1) will be evaluated according to 71-85 age group score.
4. Adequate vision, hearing, and literacy ability to allow for neuropsychological testing.
5. Able and willing to perform all study procedures.
6. Ability to provide written consent signed by the subject

Exclusion Criteria:

1. Any significant neurological condition or disorder (e.g., seizure disorder, epilepsy, brain tumors, stroke, etc.) that could cause cognitive deterioration other than suspected MCI.
2. Any medical condition or disorder that could produce cognitive deterioration (i.e., renal, respiratory, cardiac, and hepatic disease, diabetes mellitus, endocrine, metabolic or hematological disturbances) unless well controlled for at least 3 months.
3. Clinically significant abnormal serum TSH and/or B-12 and/or folic acid levels below the normal range.
4. History of any infective or inflammatory brain disease including viral, fungal or syphilitic etiologies.
5. Head trauma or injury immediately preceding cognitive deterioration, unless over 2 years have passed since full cognitive and functional recovery.
6. Depression at screening as assessed by Geriatric Depression Scale-short version (score ≥5)
7. Current suicidality at screening by Columbia Suicidality Severity Rating Scale.
8. Dementia by DSM-IV criteria.
9. Concomitant use of medications with potent psychotropic properties (e.g. antipsychotics, ADHD treatments, lithium carbonate, anti-epileptic drugs such as Gabapentin). Sedating antihistamines are allowed if administered last dose is administered at least 12 hours before cognitive testing. Usage of prescription or nonprescription antidepressant agents, lipid lowering medications, and anti-hypertensive medications with a stable dosage for more than 2 months prior study entry is permitted.
10. Concomitant use of any medications approved for the symptomatic treatment of dementia due to AD (e.g., NMDA, acetyl choline esterase inhibitors)
11. Use within 3 weeks prior to study entry of any medications with any anti-cholinergic effect (e.g. Atropine, Scopolamine, Tolterodine, Hyoscyamine, Biperiden, Benzatropine, Trihexyphenidyl, Oxybutynin).
12. Use within 4 weeks prior to the study entry of dietary supplements containing DHA, EPA, Phosphatidylserine, Phosphatidylcholine (e.g. Krill oil, Lecithin), or alpha-glycerphosphocholine (GPC).
13. Use within 4 weeks prior to the study entry of medical foods indicated for cognitive or memory impairment [e.g. Axona, Cerefolin, CerefolinNAC, Souvenaid].
14. Concomitant use of any supplements containing ingredients with nootropic or vasodilator properties (e.g., Ginkgo Biloba, Vinpocetine, Piracetam, high energy supplements).
15. Use of an investigational drug within the last 30 days.
16. Allergic reaction or sensitivity to marine products (fish/seafood) and/or soy.
17. Any known condition which in the opinion of the investigator may be possibly causing cognitive impairment other than AD (mania, alcohol or substance abuse, mental retardation, bipolar disorder, panic disorder, obsessive compulsive disorder, post-traumatic stress disorder, psychotic disorder, major psychiatric disorder preceding dementia onset or affecting brain function, major surgery ) and/or limits the successful trial completion

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 97 (Actual)
Dates: Start 2014-09; Primary Completion 2017-12-25 (Actual); Study Completion 2017-12-25 (Actual)

PRIMARY OUTCOMES:
Difference in change in the Selective Reminding Test (SRT) between the study groups. | baseline, 3, 6,12 months

SECONDARY OUTCOMES:
Mini Mental State Examination (MMSE) | baseline, 12 and 24 months
Computerized Neurological battery test (NBT) | baseline, 6, 12 and 24 months
Transition rate to dementia according to DSM-4 criteria | baseline, 3, 6, 12, 18 and 24 months
Mini Sleep Questionnaire (MSQ) | baseline, 12 and 24 months
Hamilton Anxiety Rating Scale (HAM-A). | baseline, 12 and 24 months
Selective Reminding Test (SRT) | 18 and 24 months

OTHER OUTCOMES:
Safety of phosphatidylserine versus placebo treatment | baseline, 3, 6, 12, 18 and 24 months
  Clinical laboratory safety data will be collected at baseline and 24 months. Vital signs will be measured at baseline, 12 and 24 months. Adverse events (including changes to concomitant medications) will be documented at all study visits (i.e baseline, 3, 6, 12, 18 and 24 months).

CONTACTS AND LOCATIONS:
Overall Officials: Yehudit Aharon, MD, Principal Investigator — Rambam medical center, Israel
Locations (15):
- United States (13):
  - Pharmacology Research Institute, Encino, California
  - Pharmacology Research Institute, Los Alamitos, California
  - Pharmacology Research Institute, Newport Beach, California
  - New West Physicians, PC, Golden, Colorado
  - Miami Jewish Health Systems, Miami, Florida
  - APG Research LLC, Orlando, Florida
  - University of South Florida, Tampa, Florida
  - Great Lakes Clinical Trials, Chicago, Illinois
  - Memory Enhancement Center of America, Eatontown, New Jersey
  - Princeton Medical Institute, Princeton, New Jersey
  - Integrative Clinical Trials, LLC, Brooklyn, New York
  - The Medical Research Network, New York, New York
  - Lehigh Center for Clinical Research, Allentown, Pennsylvania
- Israel (2):
  - Rambam medical center, Israel, Haifa
  - Ichilov medical center, Tel Aviv